CLINICAL TRIAL: NCT02825069
Title: Randomized Controlled Study on the Induction of Food Tolerance in Babies
Brief Title: Study on the Induction of Food Tolerance in Babies
Acronym: INTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Principal Investigator, Petri Kulmala, MD, PhD, Clinical lecturer, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Baby-INTO
Record Dates: First submitted 2016-06-28; First posted 2016-07-07 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Food Hypersensitivity
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Early introduction of solid foods starting at the age of 4 months, with foodstuff from all major groups in diet by the age of 6 months (vegetables and fruits, wheat and other grains, meat, fish, egg, dairy products). Babies presenting with mild symptoms are encouraged to continue the symptom-eliciting food.
  Interventions: Other: Early introduction of solid foods
- Control group (No Intervention): Families are advised to follow the official Finnish Nutrition Recommendations, including exclusive breastfeeding until the age of 6 months.

INTERVENTIONS:
Other: Early introduction of solid foods — Early introduction of solid foods
  Arms: Intervention group

SUMMARY:
This general population based, randomized controled trial aims at answering two major hypotheses: First, systematic early introduction of solid foods decreases the incidence of food allergy and dietary restrictions by the age of one year. Second, stimulation with the symptom-eliciting food rather than avoidance will induce tolerance in babies with non-severe allergic symptoms.

DETAILED DESCRIPTION:
All new born babies living in the city of Oulu are recruited to the study (n=1380) at their first health nurse visit (at or before 1 month of age) in the local primary care child health clinics. Families in the intervention group will get an instruction booklet including information on early systematic introduction of solid foods starting at the age of 4 months, with foodstuff from all major groups in diet by the age of 6 months (vegetables and fruits, wheat and other grains, meat, fish, egg, dairy products). Furthermore, the booklet includes information and instructions on food related symptoms and atopic eczema. Babies with mild symptoms are encouraged to continue the symptom-eliciting food. All families fill out monthly internet-based questionnaires on food diary, symptoms, diagnoses and health care visits until the age of 1 year.

ELIGIBILITY:
Inclusion Criteria:

* All newborn babies attending local Child Health Clinics

Exclusion Criteria:

* Parents unable to communicate with Finnish language (questionnaires in Finnish)

Max Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1214 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
The number of patients with dietary restrictions due to food related symptoms | By the age of one year

SECONDARY OUTCOMES:
The number of children with doctor-diagnosed food allergies | By the age of one year
The number of children with parent-reported food allergies | By the age of one year
The number of children with doctor-diagnosed atopic eczema | By the age of one year
The number of children with parent-reported atopic eczema | By the age of one year
The number of health care contacts due to food related symptoms | By the age of one year
Family experienced distress based on questionnaire | By the age of one year
  The subjective estimate of the distress (multiple choice scaled questions) related to food induced symptoms in the baby

CONTACTS AND LOCATIONS:
Overall Officials: Petri Kulmala, MD, PhD, Principal Investigator — PEDEGO-Research Unit and Medical Research Center Oulu, University of Oulu and Oulu University Hospital
Locations (1):
- PEDEGO Research Unit, University of Oulu and Oulu University Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No